CLINICAL TRIAL: NCT03803488
Title: Simulated Clinical Use Testing on the DropSafe Safety Pen Needle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HTL-Strefa S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIP v1.0 29JAN2016
Record Dates: First submitted 2019-01-09; First posted 2019-01-14 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Needle Stick
Keywords: needlestick; needlestick injury; pen needle; sharps injury prevention
MeSH Terms: conditions — Needlestick Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- simulation of injection (Experimental): The evaluator simulated the injection with the DropSafe safety pen needle and a pen injector with a sterile, water-filled cartridge using an orange.
  Interventions: Device: DropSafe safety pen needle

INTERVENTIONS:
Device: DropSafe safety pen needle

SUMMARY:
A simulated clinical use testing on the DropSafe safety pen needle

DETAILED DESCRIPTION:
This study aims to evaluate the safety of the use of DropSafe safety pen needle in the prevention of needle stick injuries (NSI) and to evaluate the user's satisfaction with regards to the handling characteristics of the product.

ELIGIBILITY:
Inclusion Criteria:

1. Minimum of age 18.
2. Able to understand and provide signed consent for the study.
3. Willing to comply with the study protocol, including being willing to answer questions and complete questionnaires.
4. Have no concerns about the ability to perform the simulated injections.
5. Have no financial interest in the sponsor (HTL-Strefa S.A.) or the MRO (NAMSA).

Exclusion Criteria:

1. If in the opinion of the sponsor or MRO, including the observer/monitor, the potential evaluator is not a good candidate for the study, including for reasons such as mental health.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-09-28 (Actual); Primary Completion 2016-12-09 (Actual); Study Completion 2016-12-09 (Actual)

PRIMARY OUTCOMES:
The true failure rate of DropSafe safety pen needle. | At time of testing, about an hour
  The failure rate of the safety feature for the DropSafe safety pen needle was estimated using the proportion of devices that fail out of the total tested. Failure was defined as NSI or contact with the needle after injection or non-complete activation of the safety feature.

SECONDARY OUTCOMES:
Ease of use | At time of testing, about an hour
  Evaluator questionnaire using five-point response scale (strongly disagree - strongly agree)
Ability to follow the instructions for use | At time of testing, about an hour
  Evaluator questionnaire using five-point response scale (strongly disagree - strongly agree)
Ease of understanding the instructions for use | At time of testing, about an hour
  Evaluator questionnaire using five-point response scale (strongly disagree - strongly agree)
Problems associated with the device | At time of testing, about an hour
  Evaluator questionnaire using five-point response scale (strongly disagree - strongly agree)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - NAMSA, Golden Valley, Minnesota
  - NAMSA, Minneapolis, Minnesota